CLINICAL TRIAL: NCT03370354
Title: The Impact of Night Nursing Activity on the Quality of Hospitalized Patients' Sleep
Brief Title: Nursing Activity and Quality of Hospitalized Patients' Sleep
Acronym: SOMACTIV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Professeur Pierre-Yves Marie, Cédric Baumann, Katie Galois, Romuald Zadra, Virginie Simon, Martine Lesny, Edith Dauchy, Saliha Sammari, Sylvie Klein (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2017-A02076-47
Record Dates: First submitted 2017-11-30; First posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Sleep Disorders, Circadian Rhythm
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: First questionnaire (spiegel questionnaire) will allow a score on 30. If the score is > 18, the patient will be in the control group.
- troubled sleeping patterns group: First questionnaire (spiegel questionnaire) will allow a score on 30. If the score is < 18, the patient will be in the troubled patterns group.
  Interventions: Behavioral: Observational

INTERVENTIONS:
Behavioral: Observational — Ask patients about sleep quality and identify reasons of troubled sleeping patterns in the units.
  Groups: troubled sleeping patterns group

SUMMARY:
This study is to determine the impact of night shift nurse's activity on patients' sleeping patterns in medical services including individual, clinical and environmental factors. The patients will be questioned in order to create both a control group and a group with troubled sleeping patterns.

DETAILED DESCRIPTION:
There are 5 speciality medical units involved. Patients must respond to the define inclusion criteria. Each patient will be asked if they agree to participate and if so will be asked to consent to participate.

Every day, nurses will give a questionnaire which will be completed by the patient to know if there were troubles sleeping patterns. If so, a second questionnaire will be completed by the patient.

Other data will be recorded such as personal informations, diagnostic, medical history, consumption habits and treatments.

The inclusion phase lasts 15 days maximum.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalize in medical units
* In the unit since one night
* Patient over 18 years old
* Patient agree to participate

Exclusion Criteria:

* Patient who can't answer to the questionnaire for health reasons
* Patient who need a specific surveillance
* Patient recently operated

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in a speciality medical units and who respond to the defined inclusion criteria. 5 units participate: nephrologye, neurology, cardiology, pneumology, endocrinology.
Sampling Method: Probability Sample
Enrollment: 328 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2019-08-15 (Estimated); Study Completion 2019-08-15 (Estimated)

PRIMARY OUTCOMES:
Presence of a sleeping disorder partially or totally related, according to patient's opinion, to night nursing activity | At the end of participation of patient- maximum at day 15 after inclusion

SECONDARY OUTCOMES:
Part of patients declaring disturbing elements related to night nursing activity | At day 15 after inclusion
  A follow up sheet is completed every day by a study nurse who asks to patient if the patient sleeps well during the previous night
Disturbing elements related to night nursing activity | Every day during 15 days
  A follow up sheet is completed every day by a study nurse who asks to patient what was the disturbing elements according to him
Individual and clinical disturbing elements | Every day during 15 days
  A follow up sheet is completed every day by a study nurse who asks to patient what was the disturbing elements according to him
Average length of patients' sleep in patients with troubled sleeping during hospitalization | Every day during 15 days
  Estimated with the Vis Morgen self administered questionnaire
Sleep quality measured by Spiegel score | Every day during 15 days
  Score from 0 to 30

CONTACTS AND LOCATIONS:
Overall Officials: Bridey Céline, Principal Investigator — CHRU Nancy France

IPD SHARING:
Plan to Share IPD: No